CLINICAL TRIAL: NCT07282132
Title: Multicenter Insights on Real-World Results Of Ropeginterferon Alpha-2B in Polycythemia Vera Patients
Brief Title: Evaluation of Real-World Data on Ropeginterferon Alfa-2b in Patients With Polycythemia Vera: Insights From a Multicenter Study
Acronym: MIRROR
Status: Not yet recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Novella Pugliese, Principal Investigator, Federico II University
Other Study IDs: AIFA-RSO-3948; AIFA-RSO-3948 (Other: A.O.U. Federico II Napoli)
Record Dates: First submitted 2025-11-26; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Polycytemia Vera
Keywords: Ropeginterferon alpha 2b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Polycythemia Vera Receiving Ropeginterferon aplha 2b: Data will be collected retrospectively from patient medical records and will include:
  1. Demographic Data
  2. Clinical Characteristics of PV
  3. Treatment Information. Details on Ropeginterferon Alfa-2b therapy: Dosage; Treatment schedule and duration; Clinical and hematologic response; Treatment discontinuation and reasons for interruption
  4. Clinical and Hematologic Response: Hematologic parameters (hemoglobin, hematocrit, platelet count, etc.); Clinical status during treatment; Spleen size assessed via abdominal ultrasound (when available); Documentation of baseline values, prior therapies, dosing schedules, and response assessments at: 3, 6, 9, 12, 18, and 24 months; Discontinuation rates and reasons for stopping therapy
  5. Molecular Response: Quantification of JAK2 V617F allele burden over time
  6. Adverse Events: Any clinically relevant complications or side effects
  Interventions: Drug: Ropeginterferon alfa-2b (BESREMi®)

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b (BESREMi®) — Ropeginterferon Alfa-2b was administered in accordance with the approved prescribing information.

SUMMARY:
This retrospective study aims to evaluate the effectiveness and safety of Ropeginterferon Alfa-2b (BESREMI) in patients with Polycythemia Vera (PV). Eligible patients have a confirmed PV diagnosis according to current criteria, have received at least one dose of Ropeginterferon, and have complete clinical and laboratory data available. The primary objective is to analyze the time course of hematologic response (complete or partial, CHR/PR) according to ELN criteria, and to identify clinical and treatment-related factors associated with achieving and maintaining response. Secondary objectives include time to response, duration of response, progression-free survival, thromboembolic event rate, safety and tolerability, treatment discontinuation, dose modifications and adherence, normalization of hematologic parameters, and changes in JAK2 V617F allele burden. Data will be collected retrospectively from medical records at participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Polycythemia Vera according to updated diagnostic criteria
* Have received at least one dose of Ropeginterferon Alfa-2b (BESREMI).
* Complete clinical and laboratory data availability for review (e.g., hematologic parameters, treatment response, adverse events).
* Followed at one of the participating study centers.
* Have signed informed consent for participation.

Exclusion Criteria:

* Have received experimental or non-approved treatments for PV during the observation period.
* Lack sufficient clinical or laboratory data to allow inclusion in the analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients diagnosed with Polycythemia Vera (PV) according to current diagnostic criteria who have received at least one administration of Ropeginterferon Alfa-2b (BESREMI) as part of their disease management. Eligible patients must have complete clinical and laboratory information available and must be followed at one of the participating centers. All participants must provide written informed consent prior to inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Analysis of Hematologic Response (CR/PR) to Ropeginterferon Alfa-2b in polycythemia vera | From enrollment to the end of treatment or at least 12 months of treatment
  Definition: Proportion of patients achieving Complete Hematologic Response (CHR) or Partial Response (PR) at each scheduled timepoint (3, 6, 9, 12, 18 and 24 months), classified according to the ELN criteria and identification of baseline and on-treatment factors associated with (a) first attainment of CHR/PR and (b) maintenance (duration) of CHR/PR.
  Assessment timepoints: Baseline, 3, 6, 9, 12, 18 and 24 months (or last available follow-up).
  Summary metrics: Proportion (%) in CHR and PR at each timepoint

SECONDARY OUTCOMES:
Time to Hematologic Response | Baseline to first documented CHR or PR (up to 24 months)
  Time (in months) from the first day of Ropeginterferon Alfa-2b treatment to achievement of CHR or PR hematologic response according to ELN criteria.
Duration of Hematologic Response | From first CHR/PR to loss or last follow-up (up to 24 months)
  Interval between first documented CHR or PR and loss of that response, death, or last follow-up.
Progression-Free Survival (PFS) | Baseline to event or last follow-up (up to 24 months)
  Time from treatment initiation to progression to post-PV myelofibrosis, acute myeloid leukemia, or death from any cause
Thromboembolic Event Rate | Baseline to last follow-up (up to 24 months)
  Proportion of patients experiencing arterial or venous thrombotic or embolic events during treatment with Ropeginterferon.
Incidence of Treatment-Emergent Adverse Events | Baseline to last follow-up (up to 24 months)
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) CTCAE v6.
Treatment Discontinuation | Baseline to last follow-up (up to 24 months)
  Proportion of patients who discontinue Ropeginterferon for adverse events, lack of efficacy, or other clinical reasons.
Dose Modifications and Adherence | Baseline to last follow-up (up to 24 months)
  Number and proportion of patients with significant dose changes (reductions or increases) and estimated adherence (planned vs observed dosing intervals).
Normalization of Hematologic Parameters | Baseline and at scheduled visits (3,6,9,12,18,24 months)
  Proportion of patients achieving target hematologic values: hematocrit <45%, leukocytes <10000/mm³, platelets <400000/mm³.
JAK2 V617F Allele Burden | Baseline and at scheduled visits (3,6,9,12,18,24 months)
  Assessment of JAK2 V617F allele burden dynamics during Ropeginterferon treatment and correlation with hematologic response.

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared to protect participant privacy and to comply with ethical and regulatory requirements.